CLINICAL TRIAL: NCT02140112
Title: A RANDOMIZED, DOUBLE-BLIND, PHASE 2A CROSSOVER STUDY TO ASSESS THE SAFETY AND EFFICACY OF TRICHURIS SUIS OVA FOR THE TREATMENT OF AUTISM SPECTRUM DISORDER
Brief Title: Efficacy and Safety of Trichuris Suis Ova (TSO) as Compared to Placebo in Autism Spectrum Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A preliminary analysis of data from this trial failed to demonstrate any signal of activity.
Sponsor: Coronado Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNDO 201-101
Record Dates: First submitted 2014-05-13; First posted 2014-05-16 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Autism
Keywords: T. suis ova; Trichuris suis ova; Autism Spectrum Disorder; ASD
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trichuris suis ova (Active Comparator): TSO 2500 x 2 doses every 2 weeks followed by TSO 7500 x 6 doses every 2 weeks
  Interventions: Biological: Trichuris suis ova
- Placebo (Placebo Comparator): Placebo 8 doses every 2 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Trichuris suis ova
  Other Names: TSO
  Arms: Trichuris suis ova
Other: Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, 2-arm, placebo-controlled crossover study in pediatric patients with autism spectrum disorder with all patients receiving 16-weeks of TSO treatment and 16 weeks of placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 5 to 17 years of age
* Patients must fulfill DSM-V diagnostic criteria for autism spectrum disorder ascertained at screening, using a clinical review confirmed by the Autism Diagnosis Observation Schedule - Second edition (ADOS-2)
* Written informed consent from parent(s) or legal guardian(s) with sufficient intellectual capacity to understand the study and support patients' adherence to the study procedures must be obtained for patients who are not emancipated. In accordance with Institutional Review Board (IRB) requirements, the patient will complete an informed assent when developmentally appropriate, to participate in the study before conduct of any study-specific procedures.
* Patients are able and willing to swallow study medication suspension.

Exclusion Criteria:

* Known diagnosis of syndromal form of Autism (e.g. Rett Syndrome, Childhood Disintegrative Disorder, Fragile X Syndrome, etc.)
* Patients who cannot discontinue anti-psychotic medication
* Patients with current active seizure disorder or who have had a seizure within the last 6 months prior to screening
* Female patient who is pregnant or breastfeeding or wishing to become pregnant during study participation or unwilling to use birth control.
* Patients who have received helminthic treatment

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2014-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Aberrant Behavior Checklist - Irritability (ABC-I) at 16 weeks | 36 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Southwest Autism Research & Resource Center, Phoenix, Arizona
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - Baber Research Group, Naperville, Illinois
  - Montefiore Medical Center Dept. of Psychiatry, Child Annex, The Bronx, New York
  - Red Oak Psychiatry, Houston, Texas